CLINICAL TRIAL: NCT05716620
Title: Utility of Abbreviated Magnetic Resonance Imaging as a Screening Tool for Hepatocellular Carcinoma in Cirrhotic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Pankaj Gupta, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: 10295
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC, cirrhosis, chronic liver disease, hepatitis B & C
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis; Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — USG and MRI will be performed on the same day. US will be performed prior to MRI. There will be two rounds of screening 6 months apart using paired US and non-enhanced AMRI.
  Other Names: USG

SUMMARY:
The goal of this study is Utility of abbrevational magnetic resonance imaging as a screening tool for hepatocellular carcinoma in cirrhotic patients.

The primary objective of the study is:

• HCC detection rate of US vs AMRI in cirrhotic patients

The secondary objective of the study are:

* False referral rate of US vs AMRI: false referral will be defined as lack of HCC on complete MRI despite a positive US or AMRI.
* Positive predictive value of US vs AMRI: The positive predictive value will be defined as the number of patients with true positive results in patients with positive US/AMRI.

Participants will be evaluated by two rounds of screening 6 months apart using paired US and non-enhanced AMRI.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common cancer and is the second leading cause of cancer related death. The most important risk factor is cirrhosis of any etiology, particularly chronic hepatitis b and hepatitis c virus infection. Curative treatment (resection, transplant, or ablation) can be offered to patients diagnosed with early HCC. As the disease remains asymptomatic, most HCCs are diagnosed at an intermediate to terminal stage. Screening is an effective strategy to diagnose early HCC. The current guidelines recommend bi-annual screening with ultrasound (US) with or without alpha- fetoprotein (AFP). The overall sensitivity for detection of HCC using US screening is 60% while it is only 22% for detection of very early and early HCC. This results in many patients having progression of HCC despite being on screening program. Although computed tomography (CT) is widely available, the cumulative radiation dose from multiple screening CT scans makes CT screening unsuitable. Magnetic resonance imaging (MRI) has a high sensitivity and specificity for diagnosis of HCC owing to its high contrast resolution. A recent study showed significantly better sensitivity of HCC detection during screening using contrast enhanced MRI (CE-MRI) as compared with US. The use of CE-MRI entails high cost and risk of nephrogenic systemic fibrosis and is not well suited for screening from the health economics standpoint. Recently abbreviated MRI (AMRI) has been proposed as an acceptable alternative to US for HCC screening. AMRI involves acquisition of only a few MRI sequences rather than the complete MRI. This results in lesser table time and in turn reduced cost. However, most of the data is from retrospective studies. We propose a prospective study to evaluate the role of AMRI for HCC screening.

ELIGIBILITY:
Inclusion Criteria:

1. Age>40 years
2. Presence of cirrhosis
3. Annual risk of HCC >5%
4. No HCC on pre-enrollment imaging not more than 6 months back.
5. Risk factors including diabetes mellitus, metabolic syndrome, family history of HCC.

Exclusion Criteria:

1. Child C status
2. Diagnosed or follow up case of HCC
3. Other malignancies
4. Pregnancy, lactation
5. Contraindications to MRI (pacemaker, cochlear implant, claustrophobia)
6. Chronic renal disease or contrast allergy precluding administration of intravenous MRI contrast agent (for reference standard)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be evaluated by two rounds of screening 6 months apart using paired US and non- enhanced AMRI. First round of screening will be performed within 6 months of a negative imaging prior to recruitment in patients who fulfill the inclusion and exclusion criteria discussed above. US and AMRI will be performed on the same day. US will be performed prior to MRI. US & AMRI will be performed by the two radiologists independently. Fasting status will not be mandatory.Radiologists will be blinded to clinical details including the risk of HCC, tumor markers and to the results of other imaging tests.
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-02-07 (Estimated); Study Completion 2025-02-07 (Estimated)

PRIMARY OUTCOMES:
HCC detection rate of US vs AMRI in cirrhotic patients | Day 7 from the time of enrolment till 12 month's scan
  number of HCCs detected by US / AMRI divided by the actual number of HCCs based reference standard

SECONDARY OUTCOMES:
False referral rate | Day 7 from the time of enrolment till 12 month's scan
  number of false positive results divided by the sum of true negative and false- positive results
Sensitivity, specificity of US vs AMRI | Day 7 from the time of enrolment till 12 month's scan
  Sensitivity, specificity of US vs AMRI
positive predictive value of US vs AMRI | Day 7 from the time of enrolment till 12 month's scan
  positive predictive value of US vs AMRI
negative predictive value of US vs AMRI | Day 7 from the time of enrolment till 12 month's scan
  negative predictive value of US vs AMRI
Survival of patients | Day 7 from the time of enrolment till 12 month's scan
  Patients who develop HCC during the 1-year follow up period using Kaplan Meier survival analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Gupta, Principal Investigator — PGIMER, CHANDIGARH
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Punjab, India

REFERENCES:
- [Background] Center MM, Jemal A. International trends in liver cancer incidence rates. Cancer Epidemiol Biomarkers Prev. 2011 Nov;20(11):2362-8. doi: 10.1158/1055-9965.EPI-11-0643. Epub 2011 Sep 15. PMID 21921256
- [Background] Kalra N, Gupta P, Chawla Y, Khandelwal N. Locoregional treatment for hepatocellular carcinoma: The best is yet to come. World J Radiol. 2015 Oct 28;7(10):306-18. doi: 10.4329/wjr.v7.i10.306. PMID 26516427
- [Background] Roayaie S, Obeidat K, Sposito C, Mariani L, Bhoori S, Pellegrinelli A, Labow D, Llovet JM, Schwartz M, Mazzaferro V. Resection of hepatocellular cancer </=2 cm: results from two Western centers. Hepatology. 2013 Apr;57(4):1426-35. doi: 10.1002/hep.25832. Epub 2013 Jan 25. PMID 22576353
- [Background] Kanwal F, Singal AG. Surveillance for Hepatocellular Carcinoma: Current Best Practice and Future Direction. Gastroenterology. 2019 Jul;157(1):54-64. doi: 10.1053/j.gastro.2019.02.049. Epub 2019 Apr 12. PMID 30986389
- [Background] Singal A, Volk ML, Waljee A, Salgia R, Higgins P, Rogers MA, Marrero JA. Meta-analysis: surveillance with ultrasound for early-stage hepatocellular carcinoma in patients with cirrhosis. Aliment Pharmacol Ther. 2009 Jul;30(1):37-47. doi: 10.1111/j.1365-2036.2009.04014.x. Epub 2009 Apr 8. PMID 19392863
- [Background] Tzartzeva K, Obi J, Rich NE, Parikh ND, Marrero JA, Yopp A, Waljee AK, Singal AG. Surveillance Imaging and Alpha Fetoprotein for Early Detection of Hepatocellular Carcinoma in Patients With Cirrhosis: A Meta-analysis. Gastroenterology. 2018 May;154(6):1706-1718.e1. doi: 10.1053/j.gastro.2018.01.064. Epub 2018 Feb 6. PMID 29425931
- [Background] Kim YK, Kim YK, Park HJ, Park MJ, Lee WJ, Choi D. Noncontrast MRI with diffusion-weighted imaging as the sole imaging modality for detecting liver malignancy in patients with high risk for hepatocellular carcinoma. Magn Reson Imaging. 2014 Jul;32(6):610-8. doi: 10.1016/j.mri.2013.12.021. Epub 2014 Jan 13. PMID 24702980
- [Background] Nakamoto A, Yamamoto K, Sakane M, Nakai G, Higashiyama A, Juri H, Yoshikawa S, Narumi Y. Reduction of the radiation dose and the amount of contrast material in hepatic dynamic CT using low tube voltage and adaptive iterative dose reduction 3-dimensional. Medicine (Baltimore). 2018 Aug;97(34):e11857. doi: 10.1097/MD.0000000000011857. PMID 30142778
- [Background] Mazhar SM, Shiehmorteza M, Kohl CA, Middleton MS, Sirlin CB. Nephrogenic systemic fibrosis in liver disease: a systematic review. J Magn Reson Imaging. 2009 Dec;30(6):1313-22. doi: 10.1002/jmri.21983. PMID 19937937